CLINICAL TRIAL: NCT07091175
Title: Singapore-Malaysian Renal Trials - Nephrotic Syndrome (SMART-NS): Dupilumab Maintenance Therapy for Steroid-dependent and Frequently Relapsing Nephrotic Syndrome
Brief Title: Dupilumab Therapy in Nephrotic Syndrome in Children
Acronym: SMART-NS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); KK Women's and Children's Hospital (Other Government); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMART-NS 01; 2024/00054 (Other: NHG DSRB, Singapore)
Record Dates: First submitted 2025-07-08; First posted 2025-07-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Nephrotic Syndrome in Children; Nephrotic Syndrome Steroid-Dependent
Keywords: Dupilumab; Steroid sensitive nephrotic syndrome; Steroid dependent nephrotic syndrome; Frequently relapsing nephrotic syndrome; Paediatric
MeSH Terms: conditions — Nephrotic Syndrome | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Parallel model with open label extension phase for participants who were randomised to placebo and relapsed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded with open label extension phase for participants who were randomised to placebo and relapsed. Participants will be randomised to receive either dupilumab or placebo. Only the designated unblinded personnel (independent of the study team) will be aware if the participant is receiving dupilumab or placebo, and draw up the correct medication into a syringe to inject into the participant. The participant, their care giver, investigators and outcomes assessor will be blinded. In the open label extension phase, there will be no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dupilumab (Experimental): Participants in the experimental arm will receive subcutaneous Dupilumab for 24 weeks at the following weight-based doses, which are identical to doses used in the treatment of atopic dermatitis (higher than that for asthma), i.e.
  * Regime A (15 to <30kg): 600mg once, then 300mg every 28 days x 5 doses.
  * Regime B (30 to <60kg): 400mg once, then 200mg every 14 days x 11 doses.
  * Regime C (60kg or more): 600mg once, then 300mg every 14 days x 11 doses.
  Interventions: Biological: Dupilumab; Drug: Co-intervention of Prednisolone wean during randomised controlled phase
- Placebo (Placebo Comparator): Participants in the control arm will receive a subcutaneous injection of matched placebo (normal saline) at the same dosing intervals as the experimental arm for 24 weeks.
  Interventions: Drug: Placebo; Drug: Co-intervention of Prednisolone wean during randomised controlled phase
- Open label extension phase (Other): On relapse, participants will be unmasked. Participants who were randomised to the placebo group will be invited to enrol into an open label extension phase. Participants will receive dupilumab in a regime identical to the experimental arm.
  Interventions: Biological: Dupilumab open label extension phase; Drug: Co-intervention of Prednisolone wean during open label extension phase

INTERVENTIONS:
Biological: Dupilumab — Subcutaneous injection of Dupilumab for 24 weeks (weight based dosing)
  Arms: Dupilumab
Drug: Placebo — Subcutaneous injection of normal saline placebo (matching dupilumab subcutaneous injection dosing) for 24 weeks
  Arms: Placebo
Drug: Co-intervention of Prednisolone wean during randomised controlled phase — The Prednisolone wean will commence 2 weeks after receiving the loading dose of Dupilumab/placebo, with each weaning step 2 weeks apart. Prednisolone will be first weaned to the same dose every other day, if the current dosing is daily (or more frequent). The dose will subsequently weaned to 4 pre-determined levels of 30mg/m2, 15mg/m2, 10mg/m2 and 5mg/m2 every other day, rounding up to the nearest 5mg. For instance, if the current dose of prednisolone is 12mg/m2 every other day, the patient will decrease the dose to 10mg/m2 every other day for 2 weeks, followed by 5mg/m2 every other day for 2 weeks, before discontinuing the drug.
  If patients enter the trial on Mycophenolate or Levamisole, this will be continued for the duration of the trial at the same dose.
  Arms: Dupilumab; Placebo
Biological: Dupilumab open label extension phase — Upon nephrotic relapse, participants will be unmasked. If they were given placebo, they will be invited to enrol in an open label extension phase to receive dupilumab for 24 weeks (with dosing identical to the experimental arm).
  Arms: Open label extension phase
Drug: Co-intervention of Prednisolone wean during open label extension phase — Patients will also receive prednisolone 60mg/m2/day as a single daily dose (max 60-80mg OD according to physician's discretion) until in remission for 3 days, before prednisolone is weaned to 40mg/m2 every other day for 2 weeks. Doses should be rounded up to nearest 5mg where possible. Prednisolone will then be weaned in steps as per the randomised controlled phase. If patients do not enter full remission after 2 weeks from enrolment into the extension phase, they will be removed from the study. Additional agents, e.g. Mycophenolate, Levamisole, Calcineurin inhibitors should not be started during this time unless there is strong clinical indication.
  Arms: Open label extension phase

SUMMARY:
The goal of this clinical trial is to learn if dupilumab works to treat severe nephrotic syndrome in children. It will also learn about the safety of dupilumab.

The main questions it aims to answer are:

* Does dupilumab reduce the time to relapse of nephrotic syndrome?
* What medical problems do participants have when taking dupilumab?

Researchers will compare dupilumab to a placebo (a look-alike substance that contains no drug) to see if dupilumab works to treat severe nephrotic syndrome.

Participants will:

* Receive an injection of dupilumab or placebo (just under the skin) every 2 weeks (if ≥30kg) or every 4 weeks (if <30kg) for 24 weeks (6 months)
* Wean down their prednisolone dose after starting the injections of dupilumab or placebo
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a nephrotic diary to record down the urine dipstick result each day, together with the dose of prednisolone taken

If protein returns in participant's urine, they will have completed the study at that point. However, if the participant is found to have received the placebo, they will be offered to receive dupilumab for up to 24 weeks.

DETAILED DESCRIPTION:
This is a multi-centre phase II double blinded randomised controlled trial which aims to assess the safety and efficacy of dupilumab for the treatment of steroid dependent or frequently relapsing steroid sensitive nephrotic syndrome in children. Participants will be randomised to receive Dupilumab or placebo via subcutaneous injection for 24 weeks. The primary efficacy end point is time to relapse. Participants who relapse will be unmasked, and if found to have received placebo, will be eligible for the open label extension phase, in which they will receive dupilumab for the following 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 years old and 18 years old at the point of recruitment with idiopathic nephrotic syndrome with disease onset between 1-18 years old
2. Steroid-dependent disease or frequently relapsing disease prior to commencement of maintenance immunosuppression
3. On oral prednisolone +/- mycophenolate or levamisole only as maintenance therapy for 6 months or more, and with inadequate disease control or steroid toxicity on therapy
4. Nephrotic relapse or partial relapse (clinical or biochemical) within the last 1 year either unprovoked or during prednisolone wean, and which responded to increase in steroids
5. In complete remission at the time of recruitment
6. Competent with, and compliant to, daily urine protein monitoring with Albustix

Exclusion Criteria:

1. Pre-existing ophthalmological conditions except refractive errors, squint or mild cataract
2. Current symptoms of helminth infection or travel to endemic areas, unless helminth infection is excluded
3. eGFR (by Bedside Schwartz equation) <60 ml/min/1.73m2
4. Received Rituximab or other B-cell depleting agents within the last 1 year
5. Biopsy proven focal segmental glomerulosclerosis
6. Known ongoing infection including HIV, Hepatitis B, Hepatitis C or tuberculosis, otherwise immunosuppressed or with frequent infections
7. Known or suspected non-compliance to medication or follow-up
8. Pregnancy or intention to become pregnant
9. Major systemic conditions, i.e. ASA Physical Status III-IV.
10. Known hypersensitivity to dupilumab or any of its excipients

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to relapse | From enrolment until date of relapse, assessed up to 24 weeks
  Relapse will be defined as either (a) urine dipstick ≥3+ on 3 consecutive days, with 1x urine protein creatinine ratio ≥200mg/mmol (2000mg/g), or (b) clinical edema in keeping with nephrotic syndrome accompanied by hypoalbuminaemia (serum albumin <30g/L), with 1x urine protein creatinine ratio ≥200mg/mmol (2000mg/g).
  Participants will be expected to record down in a nephrotic diary the urine dipstick result each day, together with the dose of prednisolone taken. Participants are expected to inform the site principal investigator (or designate) if urine dipstick is ≥3+ on 3 consecutive days, and provisions will be made for an ad-hoc urine protein creatinine ratio measurement to determine if relapse has occurred. This should be done within 24 hours of notification by participants.
  Participants will also be routinely examined for signs of nephrotic syndrome, for example edema, at study visits, and urine protein creatinine ratio will be obtained at each study visit.

SECONDARY OUTCOMES:
Time-averaged Albustix quantitation of proteinuria during study period | From enrolment until date of relapse, assessed up to 24 weeks
  Participants will be requested to record down in a nephrotic diary their urine dipstick result each day, together with the dose of prednisolone taken. The time-averaged albustix quantitation of proteinuria for the study period will then be calculated.
Minimum dose of prednisolone at the end of study | From enrolment until date of relapse, assessed up to 24 weeks
  Minimum dose of prednisolone at the end of study - at time of relapse or at 24 weeks, whichever comes first.
Percentage reduction in prednisolone dose at the end of study compared to baseline | At baseline and at time of relapse or at 24 weeks, whichever comes first
  Percentage reduction in prednisolone dose at the end of study (at time of relapse or at 24 weeks, whichever comes first) compared to baseline
Change in health-related quality of life at the end of study compared to baseline | At baseline, 1 month, 3 months, 6 months (or at time of relapse, whichever comes first)
  Health-related quality of life will be measured using the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core scales short form. There are 15 questions, where each question is scored from 0 to 4. The total score ranges from 0 to 60, where a higher score represents a lower quality of life, with more problems associated with coping with health and activities, feelings, getting along with others and work/studies.

OTHER OUTCOMES:
Change in circulating Th2 cytokines at end of study compared to baseline | At baseline, 1 month, 3 months, 6 months, (or at time of relapse, whichever comes first)
  Blood will be taken to measure for change in circulating Th2 cytokines (IL-4, IL-5, IL-13), measured in pg/ml. The required biological specimens comprise 3ml of EDTA blood and 12ml of Sodium heparin blood (or alternatively Streck Cyto-chex blood collection tube for Malaysian sites to extend sample viability). These biological specimens will require immediate priority transport to the central trial laboratory for processing on the same day (Singapore) or overnight (Malaysia).
  This is to help identify biomarkers predictive of dupilumab response.
Change in markers of Th2 polarisation at the end of study compared to baseline | At baseline, 1 month, 3 months, 6 months, (or at time of relapse, whichever comes first)
  Blood will be taken to measure for change in markers of Th2 polarisation - T-cell GATA3 (protein), STAT6 (protein) and stimulated IL-13 production, all of which will be measured as a percentage. The required biological specimens comprise 3ml of EDTA blood and 12ml of Sodium heparin blood (or alternatively Streck Cyto-chex blood collection tube for Malaysian sites to extend sample viability). These biological specimens will require immediate priority transport to the central trial laboratory for processing on the same day (Singapore) or overnight (Malaysia). This is to help identify biomarkers predictive of dupilumab response.
Number of participants with adverse events | From enrolment until date of relapse, assessed up to 24 weeks
  Adverse events would be assessed by questionnaire at each study visit every 2 weeks and reviewed by the site principal investigator within 24 hours. The following questionnaires are applicable:
  * For >17 years old, please use Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
  * For 7-17 years old, please use Pediatric-Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PED-PRO-CTCAE) if able to self-report, otherwise use Pediatric-Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (Caregiver) (PED-PRO-CTCAE [Caregiver]).
  * For <7 years old, please use Pediatric-Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (Caregiver) (PED-PRO-CTCAE [Caregiver])

CONTACTS AND LOCATIONS:
Overall Officials: Hui Kim Yap, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan CY, Teo S, Lu L, Chan YH, Lau PY, Than M, Jordan SC, Lam KP, Ng KH, Yap HK. Low regulatory T-cells: A distinct immunological subgroup in minimal change nephrotic syndrome with early relapse following rituximab therapy. Transl Res. 2021 Sep;235:48-61. doi: 10.1016/j.trsl.2021.03.019. Epub 2021 Apr 1. PMID 33812063
- [Background] Lai KW, Wei CL, Tan LK, Tan PH, Chiang GS, Lee CG, Jordan SC, Yap HK. Overexpression of interleukin-13 induces minimal-change-like nephropathy in rats. J Am Soc Nephrol. 2007 May;18(5):1476-85. doi: 10.1681/ASN.2006070710. Epub 2007 Apr 11. PMID 17429054
- [Background] Yap HK, Cheung W, Murugasu B, Sim SK, Seah CC, Jordan SC. Th1 and Th2 cytokine mRNA profiles in childhood nephrotic syndrome: evidence for increased IL-13 mRNA expression in relapse. J Am Soc Nephrol. 1999 Mar;10(3):529-37. doi: 10.1681/ASN.V103529. PMID 10073603